CLINICAL TRIAL: NCT05025384
Title: Auricular Acupressure as an Adjunct Treatment for Opioid Tapering in a Pediatric Cardiac Intensive Care Unit: A Pilot Feasibility Study
Brief Title: Jackson Pediatric Acupressure for Opioid Tapering
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Heather Jackson, Advanced Practiced Leader & Nurse Practitioner, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 210213
Record Dates: First submitted 2021-08-24; First posted 2021-08-27 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Iatrogenic Withdrawal Syndrome
MeSH Terms: interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Infants will be randomized in a 1:1 ratio to two groups - intervention vs. no intervention.
Masking Description: Participants are electronically randomized in the REDCap database.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Acupressure stickers will be applied to one ear in accordance with the NADA protocol acupuncture technique.
  Interventions: Other: Acupressure
- No Intervention (No Intervention): No intervention

INTERVENTIONS:
Other: Acupressure — Acupressure stickers will be applied to one ear in accordance with the NADA protocol acupuncture technique. Application will occur at designated points including Shen Men, Liver, and Lung: in the room with the mother; and potentially during breast feeding, holding, skin to skin contact or bottle feeds. Stickers will remain in place for 24 hours.
  At 24 hours, skin will be assessed, and stickers will then be rotated to the opposite ear every 48 - 72 hours if there are no adverse effects such as skin irritation.
  Arms: Intervention

SUMMARY:
This intervention pilot feasibility study will assess the impact of auricular acupressure as an additional non-pharmacologic therapy for infants at risk for developing Iatrogenic Withdrawal Syndrome (IWS) in the Pediatric Cardiac Intensive Care Unit (PCICU) of Monroe Carrell Jr Children's Hospital at Vanderbilt (MCJCHV). The investigators will recruit 40 healthy, 34 weeks gestational age or older infants exposed to prolonged medications (greater than 5 days) for cardiac procedures that may cause withdrawal upon cessation such as opioids, benzodiazepines, or other sedative medications. Participants will receive the auricular acupressure in addition to the standard of care such as clustered nursing care, touch, position change, environmental controls, holding, and swaddling.

DETAILED DESCRIPTION:
This intervention pilot feasibility study will assess the impact of auricular acupressure as an additional non-pharmacologic therapy for infants at risk for developing Iatrogenic Withdrawal Syndrome (IWS) in the Pediatric Cardiac Intensive Care Unit (PCICU) of Monroe Carrell Jr Children's Hospital at Vanderbilt (MCJCHV). The investigators will recruit 40 healthy, 34 weeks gestational age or older infants exposed to prolonged medications (greater than 5 days) for cardiac procedures that may cause withdrawal upon cessation such as opioids, benzodiazepines, or other sedative medications. Participants will receive the auricular acupressure in addition to the standard of care such as clustered nursing care, touch, position change, environmental controls, holding, and swaddling. Within 24 hours of implementing a weaning protocol, acupressure will be applied to three designated points of one ear following the NADA protocol acupuncture technique while also incorporating the Near-Term Infant (NTI) conceptual framework identified elements (see figure 3). Acupressure will be administered via stickers that are adhesive to the skin like a Band-Aid (see figure 1). These stickers include a vaccaria plant seed in the center that applies continuous light pressure on the designated points. This form of acupressure was selected as it is organic and does not contain metal which may interfere with emergency medical care such as imaging. After the initial 24 hours of application, stickers will be removed, the infant's skin will be assessed for any disruption such as bruising or discoloration, and the stickers will be rotated to the infant's other ear at the same NADA protocol auricular sites. Acupressure stickers will be removed and applied to the opposite ear every 48 hours until withdrawal symptoms improve (1). Withdrawal symptoms are measured every 6 hours with the enhanced Withdrawal Assessment tool (WAT) as part of the standard of care. Upon completion of the weaning regimen, infants with a score of less than or equal to 3 or less than 2 above baseline with no more than 2 rescue medication doses in 24 hours will have the acupressure removed.

ELIGIBILITY:
Inclusion Criteria:

* Infants, 34 weeks or greater gestation
* Exposure to opioids and/or benzodiazepine medications for 5 days or more
* Beginning a stable wean
* Maternal age of 18 or older

Exclusion Criteria:

* Hemodynamic instability
* Transfer to another facility prior to completion of the weaning regimen
* Death

Min Age: 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2023-01-21 (Actual); Study Completion 2023-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Jackson, MSN, APRN, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwartz L, Xiao R, Brown E, Sommers E. Auricular acupressure augmentation of standard medical management of the neonatal narcotic abstinence syndrome. Medical Acupuncture. 2011;23(3):175-86.
- [Background] Amirnovin R, Sanchez-Pinto LN, Okuhara C, Lieu P, Koh JY, Rodgers JW, Nelson LP. Implementation of a Risk-Stratified Opioid and Benzodiazepine Weaning Protocol in a Pediatric Cardiac ICU. Pediatr Crit Care Med. 2018 Nov;19(11):1024-1032. doi: 10.1097/PCC.0000000000001719. PMID 30234674
- [Background] McPherson C, Inder T. Perinatal and neonatal use of sedation and analgesia. Semin Fetal Neonatal Med. 2017 Oct;22(5):314-320. doi: 10.1016/j.siny.2017.07.007. Epub 2017 Jul 19. PMID 28734732
- [Background] Weber F, Van Beek S, Scoones G. Potential neurotoxicity of anesthetic drugs in young children: who cares? A survey among European anesthetists. Minerva Anestesiol. 2016 Mar;82(3):294-300. Epub 2015 Sep 3. PMID 26337372
- [Background] Chen X, Wan Y, Wen K, Liang T, Lin T, Li P. [Perioperative anesthetic exposure and the neurodevelopmental status of 1 year old baby underwent neonatal cardiac surgery]. Zhong Nan Da Xue Xue Bao Yi Xue Ban. 2015 Nov;40(11):1234-8. doi: 10.11817/j.issn.1672-7347.2015.11.012. Chinese. PMID 26643428
- [Background] Mebius MJ, Kooi EMW, Bilardo CM, Bos AF. Brain Injury and Neurodevelopmental Outcome in Congenital Heart Disease: A Systematic Review. Pediatrics. 2017 Jul;140(1):e20164055. doi: 10.1542/peds.2016-4055. Epub 2017 Jun 13. PMID 28607205
- [Background] Barnett AM, Machovec KA, Ames WA, Homi HM, Turi JL, Koo J, Fuller M, Jooste EH. The effect of intraoperative methadone during pediatric cardiac surgery on postoperative opioid requirements. Paediatr Anaesth. 2020 Jul;30(7):773-779. doi: 10.1111/pan.13903. Epub 2020 Jun 25. PMID 32365412
- [Background] Gupta P, Whiteside W, Sabati A, Tesoro TM, Gossett JM, Tobias JD, Roth SJ. Safety and efficacy of prolonged dexmedetomidine use in critically ill children with heart disease*. Pediatr Crit Care Med. 2012 Nov;13(6):660-6. doi: 10.1097/PCC.0b013e318253c7f1. PMID 22791093
- [Background] Edwards L, Brown LF. Nonpharmacologic Management of Neonatal Abstinence Syndrome: An Integrative Review. Neonatal Netw. 2016;35(5):305-13. doi: 10.1891/0730-0832.35.5.305. PMID 27636695
- [Background] Maguire D. Care of the infant with neonatal abstinence syndrome: strength of the evidence. J Perinat Neonatal Nurs. 2014 Jul-Sep;28(3):204-11; quiz E3-4. doi: 10.1097/JPN.0000000000000042. PMID 25062522
- [Background] Stuyt EB, Voyles CA, Bursac S. NADA Protocol for Behavioral Health. Putting Tools in the Hands of Behavioral Health Providers: The Case for Auricular Detoxification Specialists. Medicines (Basel). 2018 Feb 7;5(1):20. doi: 10.3390/medicines5010020. PMID 29414848
- [Background] Association NAD. Acupuncture Detoxification Specialist Training and Resource Manual. Fourth ed: NADA Literature Clearinghouse; 2015. 203 p.
- [Background] Bergdahl L, Berman AH, Haglund K. Patients' experience of auricular acupuncture during protracted withdrawal. J Psychiatr Ment Health Nurs. 2014 Mar;21(2):163-9. doi: 10.1111/jpm.12028. Epub 2012 Dec 12. PMID 23230968
- [Background] Landgren K, Kvorning N, Hallstrom I. Acupuncture reduces crying in infants with infantile colic: a randomised, controlled, blind clinical study. Acupunct Med. 2010 Dec;28(4):174-9. doi: 10.1136/aim.2010.002394. Epub 2010 Oct 18. PMID 20959312
- [Background] Gentry KR, McGinn KL, Kundu A, Lynn AM. Acupuncture therapy for infants: a preliminary report on reasons for consultation, feasibility, and tolerability. Paediatr Anaesth. 2012 Jul;22(7):690-5. doi: 10.1111/j.1460-9592.2011.03743.x. Epub 2011 Dec 6. PMID 22141917
- [Background] Nager AL, Kobylecka M, Pham PK, Johnson L, Gold JI. Effects of acupuncture on pain and inflammation in pediatric emergency department patients with acute appendicitis: a pilot study. J Altern Complement Med. 2015 May;21(5):269-72. doi: 10.1089/acm.2015.0024. Epub 2015 Apr 15. PMID 25875844
- [Background] Tsai SL, Reynoso E, Shin DW, Tsung JW. Acupuncture as a Nonpharmacologic Treatment for Pain in a Pediatric Emergency Department. Pediatr Emerg Care. 2021 Jul 1;37(7):e360-e366. doi: 10.1097/PEC.0000000000001619. PMID 30247457
- [Background] Yang C, Hao Z, Zhang LL, Guo Q. Efficacy and safety of acupuncture in children: an overview of systematic reviews. Pediatr Res. 2015 Aug;78(2):112-9. doi: 10.1038/pr.2015.91. Epub 2015 May 7. PMID 25950453
- [Background] Abbasoglu A, Cabioglu MT, Tugcu AU, Ince DA, Tekindal MA, Ecevit A, Tarcan A. Acupressure at BL60 and K3 Points Before Heel Lancing in Preterm Infants. Explore (NY). 2015 Sep-Oct;11(5):363-6. doi: 10.1016/j.explore.2015.07.005. Epub 2015 Jul 3. PMID 26242287
- [Background] Chen KL, Lindrea KB, Quah-Smith I, Schmolzer GM, Daly M, Schindler T, Oei JL. Magnetic noninvasive acupuncture for infant comfort (MAGNIFIC) - a single-blinded randomised controlled pilot trial. Acta Paediatr. 2017 Nov;106(11):1780-1786. doi: 10.1111/apa.14002. Epub 2017 Aug 29. PMID 28741805
- [Background] Chen LL, Su YC, Su CH, Lin HC, Kuo HW. Acupressure and meridian massage: combined effects on increasing body weight in premature infants. J Clin Nurs. 2008 May;17(9):1174-81. doi: 10.1111/j.1365-2702.2007.02147.x. PMID 18416793
- [Background] Ecevit A, Ince DA, Tarcan A, Cabioglu MT, Kurt A. Acupuncture in preterm babies during minor painful procedures. J Tradit Chin Med. 2011 Dec;31(4):308-10. doi: 10.1016/s0254-6272(12)60009-0. PMID 22462236
- [Background] Filippelli AC, White LF, Spellman LW, Broderick M, Highfield ES, Sommers E, Gardiner P. Non-Insertive Acupuncture and Neonatal Abstinence Syndrome: A Case Series from an Inner City Safety Net Hospital. Glob Adv Health Med. 2012 Sep;1(4):48-52. doi: 10.7453/gahmj.2012.1.4.007. PMID 24078899
- [Background] Raith W, Schmolzer GM, Resch B, Reiterer F, Avian A, Koestenberger M, Urlesberger B. Laser Acupuncture for Neonatal Abstinence Syndrome: A Randomized Controlled Trial. Pediatrics. 2015 Nov;136(5):876-84. doi: 10.1542/peds.2015-0676. PMID 26504123
- [Background] Raith W, Urlesberger B. Laser acupuncture as an adjuvant therapy for a neonate with neonatal abstinence syndrome (NAS) due to maternal substitution therapy: additional value of acupuncture. Acupunct Med. 2014 Dec;32(6):523-4. doi: 10.1136/acupmed-2014-010638. Epub 2014 Oct 10. No abstract available. PMID 25303949
- [Background] Jackson HJ, Lopez C, Miller S, Engelhardt B. A Scoping Review of Acupuncture as a Potential Intervention for Neonatal Abstinence Syndrome. Med Acupunct. 2019 Apr 1;31(2):69-84. doi: 10.1089/acu.2018.1323. Epub 2019 Apr 19. PMID 31031873
- [Background] Jackson HJ, Lopez C, Miller S, Englehardt B. Neonatal Abstinence Syndrome: An Integrative Review of Neonatal Acupuncture to Inform a Protocol for Adjunctive Treatment. Adv Neonatal Care. 2019 Jun;19(3):165-178. doi: 10.1097/ANC.0000000000000630. PMID 31140978
- [Background] Jackson HJ, Lopez C, Miller S, Englehardt B. Feasibility of auricular acupressure as an adjunct treatment for neonatal opioid withdrawal syndrome (NOWS). Subst Abus. 2021;42(3):348-357. doi: 10.1080/08897077.2020.1784360. Epub 2020 Jul 7. PMID 32635829
- [Background] Whelan KT, Heckmann MK, Lincoln PA, Hamilton SM. Pediatric Withdrawal Identification and Management. J Pediatr Intensive Care. 2015 Jun;4(2):73-78. doi: 10.1055/s-0035-1556749. PMID 31110855

RESULTS

PARTICIPANT FLOW:
Groups:
- Acupressure Intervention Group: Per protocol, acupressure provided.
- Control Group: Per protocol, control group.
Period: Overall Study
Arm/Group | Acupressure Intervention Group | Control Group
Started | 20 | 20
Completed | 15 | 14
Not Completed | 5 | 6
Not completed — Physician Decision | 5 | 6

BASELINE CHARACTERISTICS:
Population: 11 participants excluded per protocol and not included in analysis.
Groups:
- Intervention: Acupressure stickers will be applied to one ear in accordance with the NADA protocol acupuncture technique.
  Acupressure: Acupressure stickers will be applied to one ear in accordance with the NADA protocol acupuncture technique. Application will occur at designated points including Shen Men, Liver, and Lung: in the room with the mother; and potentially during breast feeding, holding, skin to skin contact or bottle feeds. Stickers will remain in place for 24 hours.
  At 24 hours, skin will be assessed, and stickers will then be rotated to the opposite ear every 48 - 72 hours if there are no adverse effects such as skin irritation.
- Total: Total of all reporting groups
Arm/Group | Intervention | No Intervention | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 14 | 29
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 12 | 14 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 11 | 14 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Easing of Withdrawal Symptoms as Measured by the Withdrawal Assessment Tool (WAT-1)
Description: The Withdrawal Assessment Tool- Version 1 (WAT-1) monitors opioid and benzodiazepine withdrawal symptoms in pediatric patients. A total of 19 withdrawal symptoms are rated where 0 indicates no symptoms and 10 is worst possible score in indicating intensity of withdrawal.
Time Frame: Baseline to 72 hours
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Acupressure Intervention Group | Control Group
Number analyzed (Participants) | 15 | 14
Score on a scale | 3.0 [1.5 to 4.0] | 3.0 [1.0 to 4.0]

2. Primary Outcome: Presence of Delirium as Measured by the Pediatric Confusion Assessment Method for the Intensive Care Unit (psCAM-ICU)
Description: Prevalence of Delirium will be reported using the preschool confusion assessment method for the ICU (psCAM-ICU).
  The psCAM-ICU is designed to assess for presence of delirium in critically ill children with or without mechanical ventilation. The psCAM-ICU was designed with cognitive testing that is developmentally appropriate for infants-5 years. Presence of Delirium is assessed using: 1) Acute change or fluctuating course of mental status, 2) Inattention, 3) Altered level of consciousness, 4) disorganized thinking. Presence of number 1) AND number 2) AND either number 3) OR number 4) indicates delirium is present. The following is how the data was coded: '1' for present and '2' for absent.
Time Frame: Baseline to 72 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Acupressure Intervention Group | Control Group
Number analyzed (Participants) | 15 | 14
score on a scale | 2.0 [2.0 to 2.0] | 2.0 [1.0 to 2.0]

3. Primary Outcome: Level of Sedation as Measured by the Richmond Agitation-Sedation Scale (RASS)
Description: RASS score is a 10-point scale with scores ranging from +4 (very combative, violent) to -5 (unarousable). The primary outcome was median change in RASS score between baseline (immediately before randomized intervention or standard of care) and 72 hours later.
Time Frame: Baseline to 72 hours
Measure: Median (Inter-Quartile Range); unit: score in a scale
Arm/Group | Acupressure Intervention Group | Control Group
Number analyzed (Participants) | 15 | 14
score in a scale | -0.3 [-1.0 to 0] | 0 [-0.3 to 0]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to 72 hours post intervention per the protocol
Description: Adverse event information was collected for any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research. There was one adverse event recorded in one participant.
Arm/Group | Acupressure Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 0/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acupressure Intervention Group (N=20) | Control Group (N=20)
skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — skin irritation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/84/NCT05025384/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-23): https://cdn.clinicaltrials.gov/large-docs/84/NCT05025384/ICF_001.pdf